CLINICAL TRIAL: NCT06569342
Title: Botulinum Neurotoxin Type A (BoNT-A) in Paediatric Non-neurogenic Therapy Resistant Overactive Bladder (OAB): a Cohort Study
Brief Title: Botulinum Neurotoxin Type A (BoNT-A) in Paediatric Non-neurogenic Therapy Resistant Overactive Bladder (OAB)
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Other Study IDs: OAB-BOTOX
Record Dates: First submitted 2024-08-16; First posted 2024-08-26 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Overactive Bladder; Incontinence, Daytime Urinary; Incontinence, Nighttime Urinary
MeSH Terms: conditions — Urinary Bladder, Overactive; Diurnal Enuresis; Nocturnal Enuresis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Main group: Children with OAB, who underwent intradetrusor BoNT-A-injections
  Interventions: Procedure: Intradetrusor BoNT-A

INTERVENTIONS:
Procedure: Intradetrusor BoNT-A — For intravesical injections, BoNT-A (Allergan, Irvine, CA, USA) was diluted in 0.9% saline to 10 93 international units/ml. Multiple injections were distributed throughout the detrusor, using a 94 transurethral 23-gauge injection needle under rigid cystoscopic guidance (9.8 Fr paediatric 95 cystoscope) at 10 units/kg to a maximum of 300 units. All injections were performed under general 96 anaesthesia with antibiotic prophylaxis given intra-operative as single dose intravenously.

SUMMARY:
A non-intervention cohort study on the use of Botulinum Neurotoxin Type A (BoNT-A) in Paediatric Non-neurogenic Therapy Resistant Overactive Bladder (OAB). Primary endpoint was the reduction of urinary incontinence.

DETAILED DESCRIPTION:
The investigators wanted to cunduct an analysis of children with urinary incontinence who received intradetrusor injection of BoNT-A in the period 01.01.2016 to 31.12.2020 at their centre. All patients were refractory to standard urotherapy, anticholinergics, mirabegron and combination of treatments. Patients with neurogenic bladder were excluded.

Primary endpoints were the effect on the frequency of urinary incontinence episodes. Secondary endpoints included urodynamic parameters and uroflow characteristics in relation to side effects and response to treatment.

ELIGIBILITY:
Inclusion Criteria:

* OAB
* Intradetrusor BoNT-A

Exclusion Criteria:

* Neurogenic OAB

Ages: 6 Years to 17 Years | Sex: All
Age Groups: Child
Study Population: Children refractory to standard treatment for OAB and incontinence.
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2022-01-15 (Actual); Primary Completion 2022-06-15 (Actual); Study Completion 2022-06-15 (Actual)

PRIMARY OUTCOMES:
Incontinence episodes | 1 month after treatment until request for additional treatment (up to 12 months)
  Change of incontinence episodes

SECONDARY OUTCOMES:
Response | 1 month after treatment until request for additional treatment (up to 12 months)
  Identification of predictors of response
Side effects | 1 month after treatment
  Identification of predictors of side effects

CONTACTS AND LOCATIONS:
Locations (1):
- Aarhus University Hospiral, Aarhus, Region Midt, Denmark

IPD SHARING:
Plan to Share IPD: No